CLINICAL TRIAL: NCT03867305
Title: Evaluation of the Action of MOBIDERM® on Periarticular Edema After Total Knee Prosthesis - Randomized Controlled Pilot Study
Brief Title: Evaluation of the Action of MOBIDERM® on Periarticular Edema After Total Knee Prosthesis - Randomized Controlled
Acronym: MOBŒDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IDIL/2017/SP-01
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Edema; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOBIDERM group (Experimental)
  Interventions: Device: MOBIDERM
- Control group (No Intervention)

INTERVENTIONS:
Device: MOBIDERM — Use of a MOBIDERM mobilizing band after total knee prosthesis
  Arms: MOBIDERM group

SUMMARY:
We hypothesize that the use of MOBIDERM® after total knee prosthesis allows a greater and faster resorption of periarticular edema:

* improvement of knee flexion;
* faster functional gain;
* faster decrease in postoperative pain by decreasing tissue tension.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a first total knee prosthesis (scheduled between Tuesday and Friday).
* Patient that has given his/her free and informed consent and signed the consent form.
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old (≥) and under 90 years old (<).

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study (therapeutic study)
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* The patient is allergic to latex bandages.
* The subject has contralateral amputation, pressure ulcers, severe Obstructive Arteriopathy of Lower Limbs, lymphoedema or thromboembolic event of the lower limb (ipsilateral and / or contralateral / superficial or deep or detected by postoperative Doppler).
* The subject has chronic or active wounds or any cause that hinders normal rehabilitation or the application of a bandage.
* patient with a stroke / Disabling Neurological Pathology, Chronic Immunological Pathology / Systemic Disease.
* patient with Hepatic insufficiency.
* patient with Venous insufficiency (stages 3 and 4).
* The patient is on dialysis.
* The subject has cognitive or behavioral disorders (Parkinson's disease, cerebellar syndrome, opposition, agitation, dementia).
* The subject has a history of knee surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Knee volume | Day -1
  unit: mm3
Knee volume | Day 0
  unit: mm3
Knee volume | Day 1
  unit: mm3
Knee volume | Day 5
  unit: mm3
Knee volume | Day 15
  unit: mm3
Knee volume | Month 1
  unit: mm3

SECONDARY OUTCOMES:
visual analog pain scale visual analog pain scale | Day 1
  visual scale numbered from 0 to 10 allowing patients to indicate the level of pain felt
visual analog pain scale visual analog pain scale | Day 3
  visual scale numbered from 0 to 10 allowing patients to indicate the level of pain felt
visual analog pain scale visual analog pain scale | Day 5
  visual scale numbered from 0 to 10 allowing patients to indicate the level of pain felt
visual analog pain scale visual analog pain scale | Day 15
  visual scale numbered from 0 to 10 allowing patients to indicate the level of pain felt
visual analog pain scale visual analog pain scale | Month 1
  visual scale numbered from 0 to 10 allowing patients to indicate the level of pain felt
Knee injury and Osteoarthritis Outcome (KOOS) score | day -1
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is an instrument for measuring patient-reported outcomes. It assesses short-term and long-term consequences of knee injuries and consequences of primary osteoarthritis.The KOOS has 42 elements grouped into five distinct subscales: KOOS Pain ; KOOS Symptoms; KOOS Function, daily life; KOOS Activities, sports and recreation; KOOS quality of life. The KOOS score is a percentage from 0 to 100, with 0 representing extreme problems and 100 representing no problem.
Knee injury and Osteoarthritis Outcome (KOOS) score | day 15
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is an instrument for measuring patient-reported outcomes. It assesses short-term and long-term consequences of knee injuries and consequences of primary osteoarthritis.The KOOS has 42 elements grouped into five distinct subscales: KOOS Pain ; KOOS Symptoms; KOOS Function, daily life; KOOS Activities, sports and recreation; KOOS quality of life. The KOOS score is a percentage from 0 to 100, with 0 representing extreme problems and 100 representing no problem.
Knee injury and Osteoarthritis Outcome (KOOS) score | month 1
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is an instrument for measuring patient-reported outcomes. It assesses short-term and long-term consequences of knee injuries and consequences of primary osteoarthritis.The KOOS has 42 elements grouped into five distinct subscales: KOOS Pain ; KOOS Symptoms; KOOS Function, daily life; KOOS Activities, sports and recreation; KOOS quality of life. The KOOS score is a percentage from 0 to 100, with 0 representing extreme problems and 100 representing no problem.
Measurement of knee flexion / extension | Day -1
  degree
Measurement of knee flexion / extension | Day 0
  degree
Measurement of knee flexion / extension | Day 5
  degree
Measurement of knee flexion / extension | Day 15
  degree
Measurement of knee flexion / extension | Month 1
  degree
Presence of an ecchymosis in proximity to the scar | Day 5
  Yes/no
Presence of an ecchymosis in proximity to the scar | Day 15
  Yes/no
Presence of an ecchymosis in proximity to the scar | Month 1
  Yes/no
Coloration of ecchymosis in proximity to the scar | Day 5
  Qualitative: red, pink, blue, purple, green, brown or yellow
Coloration of ecchymosis in proximity to the scar | Day 15
  Qualitative: red, pink, blue, purple, green, brown or yellow
Coloration of ecchymosis in proximity to the scar | Month 1
  Qualitative: red, pink, blue, purple, green, brown or yellow
Surface area of ecchymosis in proximity to the scar | Day 5
  Traced on OpSite Flexigrid® film: cm2
Surface area of ecchymosis in proximity to the scar | Day 15
  Traced on OpSite Flexigrid® film: cm2
Surface area of ecchymosis in proximity to the scar | Month 1
  Traced on OpSite Flexigrid® film: cm2
Resolution of the ecchymosis in proximity to the scar | Day 5
  Patient and Observer Scar Assessment Scale (observer + patient)
Resolution of the ecchymosis in proximity to the scar | Day 15
  Patient and Observer Scar Assessment Scale (observer + patient)
Resolution of the ecchymosis in proximity to the scar | Month 1
  Patient and Observer Scar Assessment Scale (observer + patient)

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, France